CLINICAL TRIAL: NCT05266612
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Biologic Effect of VG2025 as a Single Agent and in Combination Therapy With Nivolumab in Subjects With Advanced Malignant Solid Tumors
Brief Title: Phase I Study VG2025 as a Single Agent and in Combination Therapy With Nivolumab in Subjects With Advanced Malignant Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Virogin Biotech Canada Ltd (Industry)
Responsible Party: Sponsor
Organization: Virogin Biotech Ltd. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VG201-A101
Record Dates: First submitted 2022-02-09; First posted 2022-03-04 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Solid Tumor
Keywords: Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Nivolumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Monotherapy Arm (Experimental): This is an open label trial using standard 3+3 design, in up to 24 HSV seropositive subjects. This rule-based design proceeds with cohorts of three patients.
  Interventions: Drug: VG2025
- Combination Arm (Experimental): The starting dose of VG2025 in the combination cohorts will be a dose of 1.0 x108 PFU for combination cohort 1 on days 1 and 15 of every cycle. Combination cohort 2 will be dosed at 1.0 x108 PFU on Day 1 and either Day 2 or 3 in cycle 1 and 2. Day 1 only in subsequent cycles
  Interventions: Drug: VG2025; Drug: Nivolumab Injection [Opdivo]

INTERVENTIONS:
Drug: VG2025 — 1. 1.0×108PFU Day 1 and 15
  2. 2.0×108PFU Day 1 and 15
  3. 3.0×108PFU Day 1 and 15
  4. 4.0×108PFU Day 1 and 15
Drug: Nivolumab Injection [Opdivo] — Flat dose of 240 mg every two weeks.
  Arms: Combination Arm

SUMMARY:
This is a Phase 1, open-label, dose-escalation trial using standard 3+3 dose-escalation design in patients with advanced malignant solid tumors. All patients within a given dose level cohort will be treated with the same dose schedule of VG2025, administered as intratumoral injections at Day 1 and Day 15 biweekly at each treatment cycle (monotherapy cohorts 1-4 and combination cohort 1) and on day 1 and either day 2 or day 3 at the first 2 cycles followed by day 1 only at subsequent cycles (combination cohort 2). Dose limiting toxicity (DLT) evaluation period is for 4 weeks, from the start of treatment, Day 1, through Day 28.

There are two parts to this study a monotherapy arm and a combination therapy arm. In the monotherapy arm the patients will receive VG2025 only. In the combination therapy arm the patients will receive VG2025 and Nivolumab

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent.
2. Males or females aged ≥ 18 years.
3. Performance status: Eastern Cooperative Oncology Group (ECOG) 0 or 1.
4. Subject with advanced malignant solid tumors which is refractory/relapsed after and/or intolerant of standard therapies or for which no standard therapy exists or available (refer to National Comprehensive Cancer Network [NCCN] guideline).
5. At least 1 injectable cutaneous or subcutaneous lesion ≥15 mm in longest diameter and/or nodal lesions that are visible or palpable deemed injectable.
6. Seropositive for Herpes Simplex Virus (HSV).
7. Had an interval of ≥4 weeks (28 days) since exposure to immunotherapy, an interval of ≥3 weeks (21 days) since exposure to systemic chemotherapy, an interval of ≥6 weeks (42 days) since exposure to nitrosourea, and an interval of ≥4 weeks (28 days) since exposure to radiotherapy, prior to dosing.
8. Life expectancy of at least 3 months.
9. Eligibility requirements also include:

   1. Hemoglobin ≥ 90 grams (g)/liter (L),
   2. ANC ≥1.5 × 10^9/L,
10. Subjects with dermatoses without active infection will be allowed.*
11. Subjects whose baseline pulse oximetry is at least 90% on Room air.
12. Male subjects must abstain from heterosexual activities or agree to use a condom during the study and for 6 months following the end of study. Women of childbearing potential must be willing to abstain from heterosexual activities or agree to use highly effective, double-barrier contraception during the study and for 6 months following the end of study, to avoid pregnancy. Double-barrier contraception is defined as a condom AND one other form of the following:

    1. Birth control pills (The Pill)
    2. Depo or injectable birth control
    3. Intrauterine Device
    4. Birth control patch (e.g., Ortho Evra)
    5. NuvaRing®
    6. Documented evidence of surgical sterilization at least 6 months prior to the Screening visit, i.e., tubal ligation or hysterectomy for women or vasectomy for men.
13. Males must not donate sperm during the study and for at least 6 months after end of the study. Male partners of female subjects and female partners of male subjects must also use contraception, if they are of childbearing potential.
14. Females of childbearing potential must have a negative pregnancy test at Screening and on Day 1.

Exclusion Criteria:

1. Participation in any previous immunotherapy trial or any trial of any other investigational agent if half-life is more than 5 days within the last 4 weeks prior to dosing.
2. Tumors to be injected lying in mucosal regions or close to an airway, major blood vessel or spinal cord that, in the opinion of the Investigator could cause occlusion or compression in the case of tumor swelling or erosion into a major vessel in the case of necrosis.
3. Subjects with any primary Central Nervous System (CNS) malignancy including glioma and current, active, progressing CNS malignancy, including carcinomatosis meningitis are excluded. Subjects with treated brain metastases are eligible if there is no evidence of progression for at least 4 weeks after CNS-directed treatment, as ascertained by clinical examination and brain imaging (magnetic resonance imaging [MRI] or computed tomography [CT] scan) during the screening period and off systemic steroids (for at least 2 weeks prior to first dose of VG2025).
4. Major surgery within 14 days prior to Screening commencement.
5. Intercurrent serious infections within 28 days prior to Screening or treated systematically with intravenous antibiotics within 14 days prior to Screening.
6. Life-threatening illness unrelated to cancer.
7. Active Herpes or COVID-19 infections
8. Treatment with antiviral agents within 14 days prior to Screening commencement.
9. Subjects with congestive heart failure (as defined by New York Heart Association Functional Classification III or IV), unstable angina, serious uncontrolled cardiac arrhythmia, a myocardial infarction within 6 months prior to study entry or a history of myocarditis.
10. Known to test positive for human immunodeficiency virus (HIV), hepatitis B or C virus, or syphilis.
11. Subjects with a condition requiring systemic treatment with either corticosteroids (>10 milligrams (mg) daily prednisone equivalent) or other immunosuppressive medications within 14 days prior to dosing. Inhaled or topical steroids, and adrenal replacement steroid doses, are permitted in the absence of active autoimmune disease.
12. Subjects who have been on systemic anticoagulants and cannot safely hold anticoagulation for planned intratumoral injections and study procedures.
13. Subjects with prior radiation therapy to the tumor lesion to be injected are excluded from the study, unless there is evidence of tumor progression in the most recent imaging or by biopsy, following completion of radiotherapy.
14. Subjects with active or documented history of autoimmune disease within 2 years prior to Screening commencement.

    Please note that subjects with vitiligo, resolved childhood asthma/atopy, autoimmune endocrinopathy on stable replacement therapy, or psoriasis not requiring systemic treatment within the past 2 years will be allowed.
15. Subjects with history of primary immune deficiency.
16. Subjects with history of organ transplant that requires use of immunosuppressive medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-11-09 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events | 12 months
  Incidence of Adverse Events as assessed by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 5.0
MTD | 12 months
  Recommended Phase 2 Dose

SECONDARY OUTCOMES:
Level of deoxyribonucleic acid (DNA) | 12 months
  shedding profile of detectable VG2025 deoxyribonucleic acid (DNA)
interleukin level | 12 months
  evaluate the interleukin (IL)-12 and IL-15 in injected tumor (biopsy samples) and blood
ADA level of VG2025 | 12 months
  evaluate anti-drug antibody [ADA]
Nab level of VG2025 | 12 months
  evaluate neutralizing antibody [Nab]
ORR | 12 months
  Objective response rate (ORR) based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and RECIST
DoR | 12 months
  Duration of response (DoR) based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and RECIST
DCR | 12 months
  Disease control rate (DCR) based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and RECIST
PFS | 12 months
  Progression-free survival (PFS), based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and RECIST

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - MD Anderson, Houston, Texas